CLINICAL TRIAL: NCT01825421
Title: A Pilot Randomized Controlled Trial for Antibiotic Exposure in Neonatal Sepsis Using Neutrophil CD64
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding obtained
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1212011184
Record Dates: First submitted 2013-04-02; First posted 2013-04-05 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2015-07

CONDITIONS: Neonatal Early-onset Sepsis; Neonatal Late-onset Sepsis
Keywords: Infant; Infection; Newborn; Antibiotics; Neutrophil CD64; Blood Culture
MeSH Terms: conditions — Neonatal Sepsis; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (continue antibiotics) group (No Intervention): The antibiotics will be continued for at least another 24h i.e. for 48h, pending blood culture results at 48h, as per standard practice in the NICU.
- Study (discontinue antibiotics) group (Active Comparator): The intervention is to discontinue antibiotics at 24h, and he/she will be kept under observation in the NICU for at least an additional 24h, pending blood culture results at 48h.
  Interventions: Other: Intervention is to stop antibiotics at 24h .

INTERVENTIONS:
Other: Intervention is to stop antibiotics at 24h . — Stoppage of antibiotics at 24h in the intervention arm, randomization based on neutrophil CD64 values.
  Arms: Study (discontinue antibiotics) group

SUMMARY:
Unnecessary and prolonged antibiotic therapy in newborn babies can have serious consequences including development of necrotizing enterocolitis (a serious, potentially life-threatening gastrointestinal illness in premature babies), late-onset infections, resistance to antibiotics, increased length of hospital stay, and death.

Starting and continuing antibiotic therapy for blood culture-negative infections in the neonatal intensive care unit (NICU) is fairly common with numbers of such patients varying from 20%-90% of infants undergoing a sepsis evaluation in the NICU.

While blood culture results are the gold standard, there is usually a delay of up to 48-72h before the results are known. Hence, initiation and continuation of antibiotic treatment are usually based on clinical evaluation and blood count criteria which do not possess high specificity or sensitivity, and may be unreliable in the first few hours after birth or in the early stages of infection.

Since the investigators found that neutrophil CD64 (a type of protein found on the surface of a type of white blood cell that can be detected quickly in a very small amount of blood sample) has high accuracy for early detection of blood culture-proven infections in newborn babies, with extremely high negative predictive value (can identify babies definitively with no infection), the investigators will use this test to decide whether to stop or continue antibiotics in the NICU.

The investigators hypothesis is that neutrophil CD64 values can be safely used to discontinue antibiotics in newborns suspected of having infections.

The investigators aims are to utilize sequential measurements of CD64 values to stop antibiotics early in neonates being investigated for both early and late-onset infections in the NICU.

This is a prospective, randomized, controlled (RCT) trial. The study population will be derived from the sub-set of all newborn infants who have undergone investigations for presence of infection in the NICU.

ELIGIBILITY:
Inclusion Criteria:

* Infants undergoing a sepsis evaluation in the NICU

Exclusion Criteria:

* They have a major life-threatening congenital malformation
* The attending neonatologist has objections to the infant participating in the study

Ages: 1 Hour to 5 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2016-01 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Number of infants with early-onset sepsis (EOS) and late-onset sepsis (LOS) randomized to either stopping or continuing antibiotics at 24h, based on the neutrophil CD64 measurement | At 48h after initiation of antibiotics.

SECONDARY OUTCOMES:
Change in the Neutrophil CD64 Index value in neonates with/without exposure to antibiotics from 24h to 48h. | At 48h after initiation of antibiotics.

OTHER OUTCOMES:
Number of positive blood cultures in neonates from 24h to 48h with/without exposure to antibiotics. | At 48h after initiation of antibiotics.

CONTACTS AND LOCATIONS:
Locations (1):
- Yale-New Haven Children's Hospital NICU, New Haven, Connecticut, United States